CLINICAL TRIAL: NCT06903195
Title: Effect of Chokeberry Supplementation on Oxidative Stress and Gut Microbiota in Swimmers.
Brief Title: Effect of Chokeberry Supplementation on Oxidative Stress and Gut Integrity in Swimmers.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SWIMMER- SUPL
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-03

CONDITIONS: Stress Oxidative; Intestinal Permeability
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Intervention Model Description: All competitors were randomly divided into two groups (double-blind): A. supplemented (n = 12), who received two capsules with highly concentrated 18% chokeberry extract (one capsule contained 200 mg) twice a day.
  B. control (n = 10) received placebo. The supplementation period was 8 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: female swimmers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- supplemented (Experimental): The supplemented group (n=12) consumed capsules with highly concentrated 18% chokeberry extract (one capsule contained 200 mg). Each capsule also contained: chokeberry fiber, E460b magnesium salts of stearic acid (anti-caking agent), E551 silicon dioxide (anti-caking agent), hydrocypropyl methylcellulose (capsule shell) and E171 titanium dioxide (shell colour). The producer of all capsules is MLD Biotrade in Poznan.
  The swimmers took 2 capsules a day (before breakfast and dinner) for nearly 56 days (depending on length menstrual cycle phase). The swimmers sipped each capsule with glass of water.
  Interventions: Drug: Black chokeberry extract in capsules with 18% standardization of the anthocyanins content
- Placebo (Placebo Comparator): The control group (n=10) consumed capsules that were made from chokeberry fiber. The producer of all capsules is MLD Biotrade in Poznan.
  The swimmers took 2 capsules a day (before breakfast and dinner) for nearly 56 days (depending on length menstrual cycle phase). The swimmers sipped each capsule with glass of water.
  Interventions: Drug: Chokeberry fiber in capsules

INTERVENTIONS:
Drug: Black chokeberry extract in capsules with 18% standardization of the anthocyanins content — Supplement group: supplement of diet - black chokeberry extract (capsules) with 18% standardization of the anthocyanins content (one capsule contained 200 mg). Each capsule also contained: chokeberry fiber, E460b magnesium salts of stearic acid (anti-caking agent), E551 silicon dioxide (anti-caking agent), hydrocypropyl methylcellulose (capsule shell) and E171 titanium dioxide (shell colour).
  The producer of all capsules is MLD Biotrade in Poznan.
  Arms: supplemented
Drug: Chokeberry fiber in capsules — Placebo group: placebo product - chokeberry fiber (placebo capsules, which were made from chokeberry fiber).
  The producer of all capsules is MLD Biotrade in Poznan.
  Arms: Placebo

SUMMARY:
This study included 8 weeks of supplementation of black chokeberry extract with 18% standardization of the anthocyanins content (dose 2×200 mg per day) or a placebo product made from chokeberry fiber. The first research data was collected among twenty-four homogeneous female swimmers who trained intensively and attended the Sports Championship School Complex. The second research data was collected among a group of twenty-two selective and homogeneous female swimmers who attended the Sports Championship School Complex extensively.

In this study, the athletes were subjected to intensive swimming tests in breaststroke crawl (800m + 200m + 50m) with 15 minutes of active rest between test sections in the water.

Blood samples were taken from the cubital vein at three time points: before stress test (pre-exercise), one minute after the end of the test (post-exercise), and after a 3-hour recovery period (3h recovery). Measurements of morphology, 4-Hydroxynonenal (4-HNE), 8-isoprostane, cortysol, Intestinal fatty acid binding protein (I-FABP), claudin3, lipopolysaccharide (LPS), lipopolysaccharide binding protein (LBP), and levels were determined using ELISA kits (SunRed Biotechnology Company).

DETAILED DESCRIPTION:
This study included 8 weeks of supplementation of black chokeberry extract with 18% standardization of the anthocyanins content (dose 2×200 mg per day), or a placebo product made from chokeberry fiber. The first date of research completed the group of twenty-four homogeneous female swimmers, who train swimming intensively and attend the Sports Championship School Complex. The second date of research completed the group of twenty-two selective and homogeneous female swimmers, who train swimming intensively and attend the Sports Championship School Complex.

In this study, the athletes were subjected to intensive swimming tests in breaststroke crawl (800m + 200m + 50m) with 15 minutes of active rest between test sections in the water. Blood samples were taken from the cubital vein at three time points: before stress test (pre-exercise), one minute after the end of the test (post-exercise), and after a 1-hour recovery period (3h recovery).

Measurement: All determined parameters were measured with the available equipment in the ZWKF laboratory in Gorzów Wielkopolski and using commercial assay kits. Measurements were performed by the project contractors.

1. Polyethylene tubes (2.7ml) containing dipotassium ethylenediaminetetraacetic acid (EDTA) anticoagulant were used for the following tests: (a) complete blood count (7 parameters) determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland). Red blood cell indices: RBC (Red Blood Cells), HGB (Hemoglobin), HCT (Hematocrit), MCV (Mean Corpuscular Volume), MCH (Mean Corpuscular Hemoglobin), MCHC (Mean Corpuscular Hemoglobin Concentration), RDW (Red Blood Cell Distribution Width); (b) a manual blood smear was made by placing a drop of blood on a slide and then spreading it with a uniform motion. After drying, it was colored by the May Grunwald-Giemsa method according to the procedure. After drying, the stained and fixed smear was viewed under a microscope for quantitative and qualitative assessment.
2. Polyethylene clotting activator tubes (9 ml) were centrifuged to separate the morphotic elements from the serum using a centrifuge (3000 rpm for 10 min). The serum was pipetted into several Eppendorf tubes, which were then frozen (temp. -80 °C). All biochemical parameters were determined from the extracted serum: (a) using the ELISA method by the test manufacturer's instructions. The designations include the following parameters:

4-Hydroxynonenal (4-HNE), 8-isoprostane, cortysol, Intestinal fatty acid binding protein (I-FABP), claudin3, lipopolysaccharide (LPS), lipopolysaccharide binding protein (LBP).

(3) The lactate (La) concentration was determined from the capillary blood immediately after collection using a commercially available kit (Dr. Lange, Germany).

A nutritionist thoroughly analyzed the athletes' diets before each exercise test. Using a commercially available program, the amount of energy, protein, carbohydrates, fats, and fiber was then analyzed.

The experiment was conducted in accordance with the Declaration of Helsinki. The Ethical Committee of the Medical University of Poznan approved the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* valid medical examination,
* consent of the legal guardian of the underage athlete to participate in the study,
* Training experience of a minimum of three years
* Student of a sports championship school team,
* completion of the exercise test in the swimming pool - crawl style intensive test (800 m + 200 m + 50 m) on two test deadlines

Exclusion Criteria:

* antibiotic therapy,
* supplementation, use of any drugs, or oral hormonal contraceptives
* health problems within the last month

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in 4-Hydroxynonenal (4-HNE) level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of 4-Hydroxynonenal (4-HNE) [pg/ml]. ELISA method by the test manufacturer's instructions
Changes from baseline in 8-isoprostane level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of 8-isoprostane [ng/mL]. ELISA method by the test manufacturer's instructions
Changes from baseline in Cortysol level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of cortysol [ng/mL]. ELISA method by the test manufacturer's instructions
complete blood count | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Red blood cell indices: RBC (Red Blood Cells) [106 × µL-1], HGB (Hemoglobin) [g/dL] , HCT (Hematocrit) [%], MCV (Mean Corpuscular Volume)[fl], MCH (Mean Corpuscular Hemoglobin) [pg], MCHC (Mean Corpuscular Hemoglobin Concentration) [g x dL-1] , RDW (Red Blood cells Distribution Width) [%] .
a manual blood smear | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  was made by placing a drop of blood on a slide and then spreading it with a uniform motion. After drying, it was colored by the May Grunwald-Giemsa method according to the procedure. The stained and fixed smear after drying was viewed under a microscope for quantitative and qualitative assessment.
Changes from baseline in Intestinal fatty acid binfing protein (I_FABP) level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of I-FABP [pg/ml]. ELISA method by the test manufacturer's instructions
Changes from baseline in Claudin3 level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of Claudin3 [ng/ml]. ELISA method by the test manufacturer's instructions
Changes from baseline in lipopolisacharide (LPS) level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of LPS [EU/l]. ELISA method by the test manufacturer's instructions
Changes from baseline in lipopolisacharide binding protein (LBP) level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of LBP [ug/ml]. ELISA method by the test manufacturer's instructions

SECONDARY OUTCOMES:
Antropometric characteristic - height | Day 1 after overall fast
  Prior to the exercise test, the investigators measured the anthropometric parameters, including height (Seca 213 Hamburg, Deutschland) [cm]
Antropometric characteristic - weight | Day 1 after overall fast
  Prior to the exercise test, the investigators measured the anthropometric parameters, including weight (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Food record - energy | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: energy [kcal]
Food record - protein | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: protein [g]
Food record - carobhydrates | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: carobhydrates [g]
Food record - fiber | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: fiber [g]
Food record - fat | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program:: fat [g]

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No